CLINICAL TRIAL: NCT04081233
Title: The Effect of Early Stabilization of Rib Fractures on Patient-Centered Outcomes: A Randomized Clinical Trial
Brief Title: Surgical Stabilization for Rib Fractures
Acronym: SSRF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, David E. Meyer, MD, MS, FACS, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-19-0649; KL2TR003168 (NIH)
Record Dates: First submitted 2019-09-04; First posted 2019-09-09 (Actual); Results first posted 2024-02-21 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Trauma Chest; Rib Fracture Multiple
MeSH Terms: conditions — Thoracic Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early surgical stabilization (Experimental): This arm will include early surgical stabilization (within 72 hours of admission) in addition to the usual care received for patients with multiple rib fractures. Usual care will involve pain management.
  Interventions: Procedure: surgical stabilization
- Usual care (Active Comparator): This arm will be usual care only. Usual care will include pain managment.
  Interventions: Procedure: Usual care

INTERVENTIONS:
Procedure: surgical stabilization — Surgical procedure utilizing any commercially available internal rib fixation system
  Other Names: Rib plating
  Arms: Early surgical stabilization
Procedure: Usual care — Usual care typically consists of breathing exercises and pain control,often including opioids
  Arms: Usual care

SUMMARY:
The purpose of this study is to compare the usual care alone to usual care plus early surgical stabilization in adult trauma patients who have been admitted with rib fractures, to evaluate for heterogeneity of treatment effect in high risk subgroups and to determine the the impact of multiple rib fractures on post-discharge health status and time to return to work or usual physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Blunt trauma mechanism
* Severe chest wall injury (defined by one of the 3 below):

Radiographic flail segment (defined as greater than 2 fractures in greater than 3 consecutive ribs) or greater than 5 consecutive rib fractures or greater than 1 rib fractures with bicortical displacement

* At least one true rib (1-7) fractured and accessible for stabilization

Exclusion Criteria:

* Severe traumatic brain injury (best resuscitated GCS less than 8 as measured at 24 hours)
* Spinal cord injury
* Pre-existing congestive heart failure or oxygen-dependent pulmonary disease
* Any reason for which SSRF could not occur within 72 hours of admission

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2020-02-23 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David E Meyer, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Early Surgical Stabilization | Usual Care
Started | 42 | 42
Completed | 36 | 32
Not Completed | 6 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Surgical Stabilization | Usual Care | Total
Number analyzed (Participants) | 42 | 42 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (15) | 49 (15) | 49.5 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 11 | 25
  Male | 28 | 31 | 59
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Caucasian, non-Hispanic | 29 | 25 | 54
  Race/Ethnicity: Caucasian, Hispanic | 7 | 9 | 16
  Race/Ethnicity: Asian | 0 | 0 | 0
  Race/Ethnicity: Black | 6 | 7 | 13
  Race/Ethnicity: Unknown | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 42 | 42 | 84
Number of Participants Who Sustained Injury From a Motor Vehicle Collision [Count of Participants; unit: Participants] | 24 | 19 | 43
Number of Participants Who Sustained Injury From a Motorcycle Collision [Count of Participants; unit: Participants] | 7 | 5 | 12
Number of Participants Who Sustained Injury From a Fall [Count of Participants; unit: Participants] | 3 | 6 | 9
Height [Mean (Standard Deviation); unit: centimeters] | 174 (10) | 175 (10) | 174.5 (10)
Weight [Mean (Standard Deviation); unit: kilograms] | 95 (25) | 93 (22) | 94 (23.5)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 31 (6) | 30 (6) | 30.5 (6)
Emergency Department Heart Rate [Mean (Standard Deviation); unit: beats per minute] | 93 (22) | 93 (18) | 93 (20)
Emergency Department Respiratory Rate [Mean (Standard Deviation); unit: breaths per minute] | 21 (5) | 20 (5) | 20.5 (5)
Emergency Department Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 125 (30) | 127 (35) | 126 (32.5)
Emergency Department Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 79 (19) | 79 (16) | 79 (17.5)
Emergency Department Glasgow Coma Scale Score [Median (Inter-Quartile Range); unit: score on a scale] — The Glagcow Coma Scale (GCS) asses the level of consciousness in a person. The GSC is scored between 3 and 15, the higher the score the better outcome.
  score on a scale | 15 [14 to 15] | 15 [15 to 15] | 15 [14 to 15]
Injury Severity Score [Median (Inter-Quartile Range); unit: score on a scale] — The Injury Severity Score (ISS) asses the traumatic injury of 6 body regions. The total ISS score ranges between 1 to 75, a higher score indicating a worse outcome.
  score on a scale | 22 [17 to 32] | 22 [15 to 27] | 22 [17 to 29]
Abbreviated Injury Score Head [Median (Inter-Quartile Range); unit: score on a scale] — The Abbreviated Injury Scale (AIS) is an anatomically-based injury severity scoring system. The score ranges from 0 (no injury) to 6 (maximal), a higher score indicating a worse outcome.
  score on a scale | 1.5 [0 to 3] | 1 [0 to 2] | 1 [0 to 2]
Abbreviated Injury Score Face [Median (Inter-Quartile Range); unit: score on a scale] — The Abbreviated Injury Scale (AIS) is an anatomically-based injury severity scoring system. The score ranges from 0 (no injury) to 6 (maximal), a higher score indicating a worse outcome.
  score on a scale | 0 [0 to 1] | 0 [0 to 1] | 0 [0 to 1]
Abbreviated Injury Score Chest [Median (Inter-Quartile Range); unit: score on a scale] — The Abbreviated Injury Scale (AIS) is an anatomically-based injury severity scoring system. The score ranges from 0 (no injury) to 6 (maximal), a higher score indicating a worse outcome.
  score on a scale | 3 [3 to 4] | 3 [3 to 3] | 3 [3 to 4]
Abbreviated Injury Score Abdomen [Median (Inter-Quartile Range); unit: score on a scale] — The Abbreviated Injury Scale (AIS) is an anatomically-based injury severity scoring system. The score ranges from 0 (no injury) to 6 (maximal), a higher score indicating a worse outcome.
  score on a scale | 1 [0 to 2.75] | 0 [0 to 2] | 0 [0 to 2]
Abbreviated Injury Score Extremity [Median (Inter-Quartile Range); unit: score on a scale] — The Abbreviated Injury Scale (AIS) is an anatomically-based injury severity scoring system. The score ranges from 0 (no injury) to 6 (maximal), a higher score indicating a worse outcome.
  score on a scale | 2 [1 to 2] | 2 [1 to 2] | 2 [1 to 2]
Abbreviated Injury Score External [Median (Inter-Quartile Range); unit: score on a scale] — The Abbreviated Injury Scale (AIS) is an anatomically-based injury severity scoring system. The score ranges from 0 (no injury) to 6 (maximal), a higher score indicating a worse outcome.
  score on a scale | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
Number of Participants Transferred From Another Institution [Count of Participants; unit: Participants] | 15 | 19 | 34
Allocation Unit [Count of Participants; unit: Participants]
  Intensive Care | 12 | 12 | 24
  Intermediate Care | 16 | 15 | 31
  Ward | 14 | 15 | 29
Time from arrival to randomizarion [Mean (Standard Deviation); unit: hours] | 50 (22) | 54 (28) | 52 (25.1)

OUTCOME MEASURES:

1. Primary Outcome: Hospital Length of Stay
Description: Number of days patient is in the hospital
Time Frame: 180 days after admission
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Early Surgical Stabilization | Usual Care
Number analyzed (Participants) | 42 | 42
days | 9 [6 to 20] | 6 [3 to 11]

2. Secondary Outcome: Mortality
Description: Death following trauma injury involving rib fractures
Time Frame: 180 days after admission
Measure: Count of Participants; unit: Participants
Arm/Group | Early Surgical Stabilization | Usual Care
Number analyzed (Participants) | 42 | 42
Participants | 0 | 0

3. Secondary Outcome: Incidence of Respiratory Failure Requiring Mechanical Ventilation Greater Than 24 Hours
Description: number of patients who require mechanical ventilation greater than 24 hours
Time Frame: 24 hours after hospital admission
Population: Data were not collected for this outcome measure
Arm/Group | Early Surgical Stabilization | Usual Care
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Patients Requiring Tracheostomy
Description: Number of patients requiring a tracheostomy due to prolonged mechanical ventilation
Time Frame: Hospital discharge (about 20 to 30 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Early Surgical Stabilization | Usual Care
Number analyzed (Participants) | 42 | 42
Participants | 7 | 2

5. Secondary Outcome: Number of Patients Who Developed Pneumonia During the Hospitalization
Description: Number of patients diagnosed with pneumonia with greater than 10,000 cfu/ml on bronchioalveolar lavage or clinical diagnosis of pneumonia with subsequent antibiotic coverage
Time Frame: 6 months after admission
Measure: Count of Participants; unit: Participants
Arm/Group | Early Surgical Stabilization | Usual Care
Number analyzed (Participants) | 42 | 42
Participants | 9 | 5

6. Secondary Outcome: Number of Patients Who Received Regional Analgesia
Description: Number of patients utilizing regional analgesia, such as epidural, paravertebral, intercostal or serratus plane anesthesia
Time Frame: 6 months after admission
Measure: Count of Participants; unit: Participants
Arm/Group | Early Surgical Stabilization | Usual Care
Number analyzed (Participants) | 42 | 42
Participants | 7 | 3

7. Secondary Outcome: Opioid Usage
Description: Opioid usage is reported in milligrams per patient pre-randomization
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: milligrams
Arm/Group | Early Surgical Stabilization | Usual Care
Number analyzed (Participants) | 42 | 42
milligrams | 80 [50 to 167] | 79 [30 to 169]

8. Secondary Outcome: Opioid Usage
Description: Opioid usage is reported in milligrams per patient from admission to discharge
Time Frame: Hospital discharge (about 20 to 30 days)
Measure: Median (Inter-Quartile Range); unit: milligrams
Arm/Group | Early Surgical Stabilization | Usual Care
Number analyzed (Participants) | 42 | 42
milligrams
  Opioid usage (all) | 349 [218 to 686] | 177 [76 to 387]
  Opioid usage (anesthesia) | 149 [92 to 266] | 0 [0 to 90]
  Opioid usage (non-anesthesia) | 203 [89 to 477] | 125 [62 to 279]
  Daily non-anesthesia opioid exposure | 20 [9 to 43] | 19 [9 to 34]

9. Secondary Outcome: Ventilator Free Days
Description: Number of inpatient hospital days patients did not require mechanical ventilation
Time Frame: Hospital discharge (about 20 to 30 days)
Population: Data were not collected for this outcome measure.
Arm/Group | Early Surgical Stabilization | Usual Care
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Intensive Care Unit (ICU) Free Days
Description: Number of inpatient hospital days patient was not in ICU in the first 30 days
Time Frame: Hospital discharge (about 20 to 30 days)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Early Surgical Stabilization | Usual Care
Number analyzed (Participants) | 42 | 42
days | 30 [20 to 30] | 30 [29 to 30]

11. Secondary Outcome: Hospital (ICU) Free Days
Description: Number of days patient was not in the hospital during the first 30 days after admission.
Time Frame: 30 days post admission
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Early Surgical Stabilization | Usual Care
Number analyzed (Participants) | 42 | 42
days | 21 [10 to 24] | 24 [19 to 27]

12. Secondary Outcome: Re-intervention Rates for Surgical Complications
Description: The number of times a procedure was required to treat surgical complications
Time Frame: 180 days post admission
Measure: Count of Participants; unit: Participants
Arm/Group | Early Surgical Stabilization | Usual Care
Number analyzed (Participants) | 42 | 42
Participants
  Seroma | 1 | 0
  Surgical Site Infection | 1 | 0

13. Secondary Outcome: Health Status as Assessed by Visual Analog Scale (VAS) Score on the Euro Quality of Life Questionnaire (Euro QoL 5-D 5-L)
Description: Health status will be assessed by the Visual Analog Scale (VAS) Score on the Euro Quality of Life Questionnaire (Euro QoL 5-D 5-L). The Euro QoL 5-D 5-L VAS score is directly reported by participants and ranges from 0 (the worst imaginable health) to 100 (the best imaginable health). A higher score indicates a better outcome.
Time Frame: 30 days post admission
Population: Data were not collected for 5 in the early surgical stabilization arm, and data were not collected for 7 in the usual care arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Early Surgical Stabilization | Usual Care
Number analyzed (Participants) | 37 | 35
score on a scale | 65 (22) | 67 (18)

14. Secondary Outcome: Health Status as Assessed by Visual Analog Scale (VAS) Score on the Euro Quality of Life Questionnaire (Euro QoL 5-D 5-L)
Description: as for outcome 13
Time Frame: 90 days post admission
Population: Data were not collected for 8 in the early surgical stabilization arm, and data were not collected for 10 in the usual care arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Early Surgical Stabilization | Usual Care
Number analyzed (Participants) | 34 | 32
score on a scale | 69 (24) | 73 (23)

15. Secondary Outcome: Health Status as Assessed by Visual Analog Scale (VAS) Score on the Euro Quality of Life Questionnaire (Euro QoL 5-D 5-L)
Description: as for outcome 13
Time Frame: 180 days post admission
Population: Data were not collected for 6 in the early surgical stabilization arm, and data were not collected for 10 in the usual care arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Early Surgical Stabilization | Usual Care
Number analyzed (Participants) | 36 | 32
score on a scale | 74 (23) | 77 (20)

16. Secondary Outcome: Health Status as Assessed by Index Score on the Euroqol-5D-5L
Description: Health Status will be assessed by the index score on the Euro Quality of Life Questionnaire (Euro QoL 5-D 5-L). The Euro QoL 5-D 5-L index score ranges from 0 (a state as bad as being dead) to 1 (full health), and it is a summary score based on societal preference weights for the cumulative health states measured by 5 different dimensions (Mobility, Self-care, Daily activities, Pain/Discomfort, Anxiety/ Depression). It is calculated using the 2017 United States time trade-off valuation data set. A higher score indicates a better outcome.
Time Frame: 30 days post admission
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Early Surgical Stabilization | Usual Care
Number analyzed (Participants) | 37 | 35
score on a scale | 0.44 (0.34) | 0.53 (0.27)

17. Secondary Outcome: Health Status as Assessed by Index Score on the Euroqol-5D-5L
Description: as for outcome 16
Time Frame: 90 days post admission
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Early Surgical Stabilization | Usual Care
Number analyzed (Participants) | 34 | 32
score on a scale | 0.56 (0.32) | 0.61 (0.36)

18. Secondary Outcome: Health Status as Assessed by Index Score on the Euroqol-5D-5L
Description: as for outcome 16
Time Frame: 180 days post admission
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Early Surgical Stabilization | Usual Care
Number analyzed (Participants) | 36 | 32
score on a scale | 0.69 (0.32) | 0.77 (0.26)

19. Secondary Outcome: Health Status as Indicated by Level of Impairment as Assessed by the Euroqol-5D-5L
Description: Level of impairment will be assessed for five dimensions (Mobility, Self-care, Daily activities, Pain, Anxiety) by using the Euro Quality of Life Questionnaire (Euro QoL 5-D 5-L). Each dimension is rated at five levels: no impairment (1); minor impairment (2); moderate impairment (3); severe impairment (4); and extreme impairment (5). A higher score indicates a worse outcome.
Time Frame: 30 days post admission
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Early Surgical Stabilization | Usual Care
Number analyzed (Participants) | 37 | 35
score on a scale
  Mobility | 3 [2 to 3] | 2 [1 to 2]
  Self-care | 2 [2 to 3] | 2 [1 to 2]
  Usual activities | 3 [2 to 5] | 3 [2.5 to 5]
  Pain | 3 [2 to 3] | 3 [2 to 3]
  Anxiety | 2 [1 to 3] | 2 [1 to 3]

20. Secondary Outcome: Health Status as Indicated by Level of Impairment as Assessed by the Euroqol-5D-5L
Description: Level of impairment will be assessed for five dimensions (Mobility, Self-care, Daily activities, Pain/Discomfort, Anxiety/ Depression) by using the Euro Quality of Life Questionnaire (Euro QoL 5-D 5-L). Each dimension is rated at five levels: no impairment (1); minor impairment (2); moderate impairment (3); severe impairment (4); and extreme impairment (5). A higher score indicates a worse outcome.
Time Frame: 90 days post admission
Population: as for outcome 14
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Early Surgical Stabilization | Usual Care
Number analyzed (Participants) | 34 | 32
score on a scale
  Mobility | 2 [1 to 3] | 1 [1 to 3]
  Self-care | 1 [1 to 2.5] | 1 [1 to 3]
  Usual activities | 3 [2 to 3] | 2 [1 to 3.25]
  Pain | 3 [2 to 3] | 2 [2 to 3]
  Anxiety | 2 [1 to 3] | 2 [1 to 2]

21. Secondary Outcome: Health Status as Indicated by Level of Impairment as Assessed by the Euroqol-5D-5L
Description: as for outcome 20
Time Frame: 180 days post admission
Population: as for outcome 15
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Early Surgical Stabilization | Usual Care
Number analyzed (Participants) | 36 | 32
score on a scale
  Mobility | 1 [1 to 2] | 1 [1 to 2]
  Self-care | 1 [1 to 1] | 1 [1 to 1]
  Usual activities | 2 [1 to 3] | 1.5 [1 to 3]
  Pain | 2 [2 to 3] | 2 [1 to 3]
  Anxiety | 1 [1 to 2] | 1 [1 to 2]

22. Secondary Outcome: Time From Injury to Return to Work
Description: Number of days from time of injury until patient was able to return to work prior to injury per patient's assessment
Time Frame: 180 days post admission
Population: as for outcome 15
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Early Surgical Stabilization | Usual Care
Number analyzed (Participants) | 36 | 32
days | 48 [35 to 89] | 43 [35 to 55]

23. Secondary Outcome: Time From Injury to Resolution of Pain
Description: Number of days from time of injury to time patient verbalized pain was resolved
Time Frame: 180 days post admission
Population: as for outcome 15
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Early Surgical Stabilization | Usual Care
Number analyzed (Participants) | 36 | 32
days | 76 [35 to 104] | 54 [25 to 73]

24. Secondary Outcome: Time From Injury to Return to Usual Activity
Description: Number of days from time of injury until patient was able to return to usual activities prior to injury per patient's assessment
Time Frame: 180 days post admission
Population: as for outcome 15
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Early Surgical Stabilization | Usual Care
Number analyzed (Participants) | 36 | 32
days | 92 [77 to 119] | 67 [52 to 112]

25. Secondary Outcome: Number of Participants Prescribed Opioids at Discharge
Time Frame: Hospital discharge (about 20 to 30 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Early Surgical Stabilization | Usual Care
Number analyzed (Participants) | 42 | 42
Participants
  Tramadol | 22 | 24
  Other Opioid | 3 | 4

26. Secondary Outcome: Number of Participants Back to Work or Normal Physical Activity
Time Frame: 30 days post admission
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Early Surgical Stabilization | Usual Care
Number analyzed (Participants) | 37 | 35
Participants | 5 | 5

27. Secondary Outcome: Number of Participants Back to Work or Normal Physical Activity
Time Frame: 90 days post admission
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Early Surgical Stabilization | Usual Care
Number analyzed (Participants) | 34 | 32
Participants | 14 | 17

28. Secondary Outcome: Number of Participants Back to Work or Normal Physical Activity
Time Frame: 180 days post admission
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Early Surgical Stabilization | Usual Care
Number analyzed (Participants) | 36 | 32
Participants | 19 | 19

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Early Surgical Stabilization | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/42
Serious Adverse Events (participants affected / at risk) | 12/42 | 8/42
Other Adverse Events (participants affected / at risk) | 6/42 | 2/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Early Surgical Stabilization (N=42) | Usual Care (N=42)
Surgical site infection (Injury, poisoning and procedural complications) | 1 | 0 — Participants in the usual care arm are not at risk for the surgical complication of surgical site infection.
Deep vein Thrombosis (Vascular disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 9 | 5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Early Surgical Stabilization (N=42) | Usual Care (N=42)
Seroma (Injury, poisoning and procedural complications) | 1 | 0 — Participants in the usual care arm are not at risk for the surgical complication of seroma.
Retained Hemothorax (Injury, poisoning and procedural complications) | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-28): https://cdn.clinicaltrials.gov/large-docs/33/NCT04081233/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-12): https://cdn.clinicaltrials.gov/large-docs/33/NCT04081233/ICF_001.pdf